CLINICAL TRIAL: NCT01682239
Title: Effects of Different Right Ventricular Lead Positioning on Cardiac Contraction Measured by Cardiac MRI: a Pilot Trial
Brief Title: Effects of Right Ventricular Pacemaker Lead Position Assessed by MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alfred A Kocher, MD, MD., Prof., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EC 023/2012
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Late Complication From Cardiac Pacemaker Implantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RVAP lead (Experimental): Pacemaker lead implantation:
  Pacemaker leads will be placed in specific predefined RA and RV sites according to randomization. In this arm pacemaker leads will be placed in the RV apex. The successful lead positioning at its target location will be verified by surface ECG and by fluoroscopy.
  Interventions: Other: RVAP
- RVSP arm (Experimental): Pacemaker lead implantation:
  Pacemaker leads will be placed in specific predefined RA and RV sites according to randomization. In this arm pacemaker leads will be placed in the RV septum. The successful lead positioning at its target location will be verified by surface ECG and by fluoroscopy.
  Interventions: Other: RVSP

INTERVENTIONS:
Other: RVAP — In this arm pacemaker leads will be placed in the RV apex.
  Arms: RVAP lead
Other: RVSP — In this arm pacemaker leads will be placed in the RV septum.
  Arms: RVSP arm

SUMMARY:
Chronic right ventricular apical pacing has been associated with negative hemodynamic effects. Clinical outcome of right ventricular pacing can be influenced by multiple factors. An important factor seems to be optimal lead positioning. Data regarding left ventricular function impaired by lead positioning is insufficient. The aim of the present study therefore is to compare right ventricular apical pacing (RVAP) with right ventricular septal pacing (RVSP). Outcome measurements are echocardiographic features, magnetic resonance imaging and clinical outcome.

ELIGIBILITY:
Inclusion criteria:

* patients with dysrhythmia requiring dual-chamber pacemaker implantation
* planed MRI-pacemaker implantation (Accent MRI System,St. Jude Medical)
* age between 18-90 years
* no absolute pacemaker dependence
* no present heart failure or any significant coronary heart disease (exclusion by anamnesis and echocardiography - LVH <15mm, LV EF>50%)
* no previous myocardial infarction or significant coronary artery disease
* life expectancy > 1 year
* patients willing to participate in follow-up

Exclusion criteria:

* Contraindications for MRI (Brain aneurysm clips, artificial heart valves, artificial joints, vascular stents)
* Any contraindication for surgery
* Absolute pacemaker dependence
* Claustrophobia
* GFR<30ml/min/1,73m2
* Allergy to contrast agent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Ejection Fraction | 6 month
  As primary endpoint the difference of ventricular function in both groups will be taken. Therefore the Ejection Fraction is measured in cardiac MRI and Echocardiography. There may be a different development of contraction, whether the lead is placed in the ventricular apex or the ventricular septum.

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Kocher, MD, Principal Investigator — Department of Cardiac Surgery
Locations (1):
- Department of Cardiac Surgery, MUV, Vienna, Vienna, Austria

REFERENCES:
- [Background] Beinart R, Nazarian S. MRI-Conditional Cardiac Implantable Electronic Devices: What's New and What Can We Expect in the Future? Curr Treat Options Cardiovasc Med. 2012 Oct;14(5):558-64. doi: 10.1007/s11936-012-0197-2. PMID 22851216
- [Background] Cano O, Osca J, Sancho-Tello MJ, Sanchez JM, Ortiz V, Castro JE, Salvador A, Olague J. Comparison of effectiveness of right ventricular septal pacing versus right ventricular apical pacing. Am J Cardiol. 2010 May 15;105(10):1426-32. doi: 10.1016/j.amjcard.2010.01.004. Epub 2010 Mar 30. PMID 20451689
- [Background] Inoue K, Okayama H, Nishimura K, Saito M, Yoshii T, Hiasa G, Sumimoto T, Inaba S, Suzuki J, Ogimoto A, Funada J, Higaki J. Right ventricular septal pacing preserves global left ventricular longitudinal function in comparison with apical pacing: analysis of speckle tracking echocardiography. Circ J. 2011;75(7):1609-15. doi: 10.1253/circj.cj-10-1138. Epub 2011 May 20. PMID 21597204